CLINICAL TRIAL: NCT04401033
Title: Prospective Observational Study Evaluating the Increased Risk of SARS-CoronaVirus-2 (SARS-CoV-2) Infection Associated With Endoscopic Procedures (DECORE Study)
Brief Title: Increased Risk of SARS-CoronaVirus-2 (SARS-CoV-2) Infection Associated With Endoscopy (DECORE Study)
Acronym: DECORE
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal co-investigator, Hospital del Rio Hortega
Other Study IDs: 003
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV 2; COVID
Keywords: COVID; SARS-CoV 2; Endoscopy
MeSH Terms: interventions — Endoscopy, Gastrointestinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Endoscopic cohort: Endoscopic examinations: They will be carried out according to the recommendations of the Spanish society for digestive endoscopy (SEED). In summary, the patient will perform a hand wash with hydroalcoholic solution before entering the endoscopy room, and will put on a surgical mask and gloves. Personnel close to the patient will wear an FFP2 mask, exceptionally a surgical mask, a gown (waterproof in high-risk examinations as established in the SEED guidelines), a cap, nitrile gloves and face shield or safety glasses (reusable) and shoe covers. The examinations will be performed by endoscopist-guided sedation in accordance with current clinical guidelines.
  Interventions: Procedure: Gastrointestinal endoscopy
- Ultrasonography cohort: Abdominal ultrasound: They will be carried out according to international clinical guidelines (12). The explorer will wear an FFP2 mask, exceptionally a surgical mask, a gown, a hat, nitrile gloves, and a face shield or safety glasses (reusable) and shoe covers. The gel bottle, transducer, and stretcher will be washed prior to each scan with low-level disinfectant
  Interventions: Procedure: Abdominal ultrasound
- Telephonic cohort: The patient will be telephonically contacted for a medical visit.
  Interventions: Behavioral: Telephonic medical visit

INTERVENTIONS:
Behavioral: Telephonic medical visit — The patient will receive a telephonic call passing a medical visit
  Groups: Telephonic cohort
Procedure: Gastrointestinal endoscopy — Upper or lower GI endoscopy according to clinical practice and current guidelines
  Groups: Endoscopic cohort
Procedure: Abdominal ultrasound — Diagnostic abdominal ultrasound according to the current guidelines
  Groups: Ultrasonography cohort

SUMMARY:
The aim of our study to compare the proportion of patients who develop SARS-CoV-2 disease in 3 groups: patients undergoing a abdominal ultrasound examination in a Specialty Center, patients undergoing endoscopic procedure in a third level hospital with CoronaVirus Disease (COVID-19) hospitalization plants and patients who make a telephonic visit (do not go to the hospital) in the digestive system service.

DETAILED DESCRIPTION:
Patients will undergo a telephonic interview 48-96h before the procedure where will ask about the presence of symptoms suggestive of SARS-CoV-2 infection. Optionally, they will also be carried out a scan (PCR) to detect infection 48-96h before procedure, withdrawing from the study patients with positive PCR or infection suspected by clinical data according to the questionnaire, after evaluating the responses to the questionnaire by one of the members of the research team.

Endoscopic examinations will be carried out according to the recommendations of the Spanish Society for Digestive Endoscopy (SEED). The patient will perform a hand wash with solution hydroalcoholic before entering the endoscopy room, and you will be placed a surgical mask and gloves. Staff close to the patient will carry FFP2 mask, exceptionally surgical mask, gown (waterproof in high-risk examinations as established in the SEED guidelines), hat, nitrile gloves and face shield or safety glasses (reusable) and shim covers. The examinations will be carried out using sedation guided by endoscopist according to current clinical guidelines.

Ultrasonographic examinations (US) will be carried out according to clinical guideline. The examinator will wear a filtering face pieces 2 (FFP2) mask, exceptionally surgical mask, gown, cap, nitrile gloves and face shield or goggles safety (reusable) and shoe covers. The gel bottle, the transducer and the gurney will be washed before each US with low level disinfectant.

Patients who meet the inclusion criteria and do not have any exclusion criteria will be invited to participate in the study. The patients who agree to participate will complete the informed consent according to the law 41/2002 of patient autonomy without for that reason alter the relationship with your doctor or cause any harm to your treatment. The monitoring period will have a maximum duration of 17 days. It will consist of a telephone control through a pre-established checklist. In case of any positive answer to the questionnaire, it will be completed the study through the consultation of the investigators by means of a polymerase chain reaction (PCR).

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for an ambulatory endoscopy, an ambulatory abdominal ultrasound, or a telephonic visit Age younger than 18 years.

Exclusion criteria:

Refusal to sign the informed consent Immunosuppression (steroid treatment with a dose of 20 mg or more of prednisone daily, azathioprine, cyclosporine, mercaptopurine, methotrexate, mycophenolate, tacrolimus, everolimus, chemotherapeutic agents, anti-tumoral necrosis factor (TNF)-α drugs or other biological treatments for inflammatory bowel disease) Immunodeficiency due to a non-pharmacological cause (HIV, hematological dyscrasias, primary immunodeficiencies ...) Previous confirmed diagnosis (by PCR or serology) of SARS-CoV-2 disease. Diagnosis of previous suspicion (documented in the medical history by a physician) of SARS-CoV-2 disease.

Previous clinical picture compatible with SARS-CoV-2 in the previous 2 months (defined as any positive response to the check-list questionnaire contained in Annex III) Cognitive impairment or hearing impairment preventing the phone visit Habitual residence outside the province of Valladolid Ultrasound interventionism (liver biopsy, ultrasound-guided paracentesis, biliary drainage ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for an ambulatory endoscopy, an ambulatory abdominal ultrasound, or a telephonic visit
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection in patients | may-june 2020
  Proportion of patients who develop SARS-CoV-2 infection in 3 groups: patients undergoing an abdominal ultrasound examination in a Specialty Center, patients undergoing an endoscopic examination in a third-level hospital with hospitalization facilities COVID-19 and patients who make a non-face-to-face consultation (do not go to the hospital) in the digestive system service

SECONDARY OUTCOMES:
SARS-CoV-2 infection in HCW | may-june 2020
  Number of Health Care Workers (HCW) who develop SARS-CoV-2 infection in endoscopy service in this period

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sociedad Espanola de Patologia Digestiva; Asociacion Espanola de Gastroenterologia. Recommendations by the SEPD and AEG, both in general and on the operation of gastrointestinal endoscopy and gastroenterology units, concerning the current SARS-CoV-2 pandemic (March, 18). Rev Esp Enferm Dig. 2020 Apr;112(4):319-322. doi: 10.17235/reed.2020.7052/2020. PMID 32202911
- [Background] Huh S. How to train health personnel to protect themselves from SARS-CoV-2 (novel coronavirus) infection when caring for a patient or suspected case. J Educ Eval Health Prof. 2020 Jan;17:10. doi: 10.3352/jeehp.2020.17.10. Epub 2020 Mar 7. No abstract available. PMID 32150796
- [Background] Liu Z, Zhang Y, Wang X, Zhang D, Diao D, Chandramohan K, Booth CM. Recommendations for Surgery During the Novel Coronavirus (COVID-19) Epidemic. Indian J Surg. 2020 Apr;82(2):124-128. doi: 10.1007/s12262-020-02173-3. Epub 2020 Apr 11. PMID 32292252
- [Background] The Lancet. COVID-19: protecting health-care workers. Lancet. 2020 Mar 21;395(10228):922. doi: 10.1016/S0140-6736(20)30644-9. No abstract available. PMID 32199474
- [Background] Hunter E, Price DA, Murphy E, Schim van der Loeff I, Baker KF, Lendrem D, Lendrem C, Schmid ML, Pareja-Cebrian L, Welch A, Payne BAI, Duncan CJA. First experience of COVID-19 screening of health-care workers in England. Lancet. 2020 May 2;395(10234):e77-e78. doi: 10.1016/S0140-6736(20)30970-3. Epub 2020 Apr 22. No abstract available. PMID 32333843
- [Background] Chow EJ, Schwartz NG, Tobolowsky FA, Zacks RLT, Huntington-Frazier M, Reddy SC, Rao AK. Symptom Screening at Illness Onset of Health Care Personnel With SARS-CoV-2 Infection in King County, Washington. JAMA. 2020 May 26;323(20):2087-2089. doi: 10.1001/jama.2020.6637. PMID 32301962
- [Background] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930
- [Background] Nishiura H, Kobayashi T, Miyama T, Suzuki A, Jung SM, Hayashi K, Kinoshita R, Yang Y, Yuan B, Akhmetzhanov AR, Linton NM. Estimation of the asymptomatic ratio of novel coronavirus infections (COVID-19). Int J Infect Dis. 2020 May;94:154-155. doi: 10.1016/j.ijid.2020.03.020. Epub 2020 Mar 14. No abstract available. PMID 32179137
- [Background] Day M. Covid-19: identifying and isolating asymptomatic people helped eliminate virus in Italian village. BMJ. 2020 Mar 23;368:m1165. doi: 10.1136/bmj.m1165. No abstract available. PMID 32205334
- [Background] van Doremalen N, Bushmaker T, Morris DH, Holbrook MG, Gamble A, Williamson BN, Tamin A, Harcourt JL, Thornburg NJ, Gerber SI, Lloyd-Smith JO, de Wit E, Munster VJ. Aerosol and Surface Stability of SARS-CoV-2 as Compared with SARS-CoV-1. N Engl J Med. 2020 Apr 16;382(16):1564-1567. doi: 10.1056/NEJMc2004973. Epub 2020 Mar 17. No abstract available. PMID 32182409
- [Background] World Federation for Ultrasound in Medicine and Biology Safety Committee (Jacques S. Abramowicz, Iwaki Akiyama, David Evans, J. Brian Fowlkes, Karel Marsal, Yusef Sayeed and Gail ter Haar); Abramowicz JS, Basseal JM. World Federation for Ultrasound in Medicine and Biology Position Statement: How to Perform a Safe Ultrasound Examination and Clean Equipment in the Context of COVID-19. Ultrasound Med Biol. 2020 Jul;46(7):1821-1826. doi: 10.1016/j.ultrasmedbio.2020.03.033. Epub 2020 Apr 4. No abstract available. PMID 32327199
- [Background] Repici A, Aragona G, Cengia G, Cantu P, Spadaccini M, Maselli R, Carrara S, Anderloni A, Fugazza A, Pace F, Rosch T; ITALIAN GI-COVID19 Working Group. Low risk of COVID-19 transmission in GI endoscopy. Gut. 2020 Nov;69(11):1925-1927. doi: 10.1136/gutjnl-2020-321341. Epub 2020 Apr 22. No abstract available. PMID 32321857

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/33/NCT04401033/Prot_SAP_000.pdf